CLINICAL TRIAL: NCT01855555
Title: The Incidence and Nature of Adverse Events During Pediatric Sedation for MRI/CT in One Korean University Hospital: Prospective Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0688
Record Dates: First submitted 2013-05-09; First posted 2013-05-16 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Children Requiring Sedation for MRI/CT
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sedation group: Children requiring sedation for MRI/CT
  Interventions: Drug: sedation with propofol

INTERVENTIONS:
Drug: sedation with propofol — When a patient is admitted to the Pediatric Sedation Center, a presedation assessment is performed by hospitalists. Then Pediatric sedation is performed by protocol in the sedation unit.
  Data on demographics, primary illness, ASA, snoring history, URI symptom, medications used, procedure and recovery times, medication doses, outcomes of anesthesia, airway interventions and adverse events will be reported.

SUMMARY:
Sedation and anesthesia for which to perform diagnostic imaging represents a rapidly growing field of practice, especially in children. Propofol is the most common sedative drug administered for MRI/CT. However, this drug is associated with adverse events, including pulmonary complications, and there has been no report on these complications in Korea. In this prospective observation study, the investigators will report the nature and frequency of adverse events associated with propofol-based sedation for MRI/CT.

ELIGIBILITY:
Inclusion Criteria:

* Requiring sedation for MRI/CT, aged 0- 18 years

Exclusion Criteria:

* Parent refusal of participation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children requiring sedation for MRI/CT
Sampling Method: Non-Probability Sample
Enrollment: 2948 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 24 hours
  The investigators will record all adverse events that are associated with pediatric sedation for MRI/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Cravero JP, Beach ML, Blike GT, Gallagher SM, Hertzog JH; Pediatric Sedation Research Consortium. The incidence and nature of adverse events during pediatric sedation/anesthesia with propofol for procedures outside the operating room: a report from the Pediatric Sedation Research Consortium. Anesth Analg. 2009 Mar;108(3):795-804. doi: 10.1213/ane.0b013e31818fc334. PMID 19224786